CLINICAL TRIAL: NCT07266142
Title: Prospective Collection of Clinical Data and Human Body Material (HBM): Blood (Serum, Plasma, DNA) and Tissue of Cutaneous Melanoma and Non Melanoma Patients. Biobank Huidkanker
Brief Title: Prospective Collection of Clinical Data and Human Body Material (HBM) of Cutaneous Melanoma and Non Melanoma Patients. Biobank Huidkanker
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S70567
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Skin Cancer, Non-Melanoma; Skin Cancer Melanoma
Keywords: Prospective Collection; Skin Cancer; Human Body Material
MeSH Terms: conditions — Skin Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (serum, plasma) and tissue samples (tumor and adjacent normal skin).
  Samples will be stored long-term in the UZ Leuven Biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biobank Collection Arm: Participants diagnosed with cutaneous melanoma or non-melanoma skin cancer will provide informed consent for collection and long-term storage of human body material (HBM)-blood (serum, plasma, DNA) and tissue-and associated clinical data for future research.
  Interventions: Other: Collection of Human Body Material and Clinical Data

INTERVENTIONS:
Other: Collection of Human Body Material and Clinical Data — Blood sampling (serum, plasma, DNA) Tissue sampling (additional biopsy if consented) Completion of Cancer Worry Scale questionnaire

SUMMARY:
The goal of this clinical trial is to set up a prospective, fit-for-purpose collection of human body material (HBM)-blood (serum, plasma, DNA) and tissue-and standardized clinical data of patients with cutaneous melanoma and non-melanoma skin cancer.

The main questions it aims to answer are:

* To create a biobank with samples of human body material (HBM): blood (serum/plasma/DNA) and tissue and clinical data of patients with cutaneous melanoma and non-melanoma.
* To support future research questions (after specific approval of the Ethics Committee) by using the biobank (through satellite protocols).

If there is a comparison group: Not applicable (umbrella protocol for collection only).

Participants will:

* Share demographics, medical and surgical history, risk factors.
* Complete Cancer Worry Scale questionnaire.
* Provide biological samples:

  * Blood samples (serum, plasma, DNA).
  * Tissue samples (residual tissue or additional biopsy if consented).

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
* Adult subjects (>18 years of age) at time of enrolment.
* Subjects diagnosed with cutaneous melanoma or Non-melanoma skin cancer.
* Adult subjects able and willing to provide informed consent.

Exclusion Criteria:

* Subjects unable or not willing to provide informed consent.
* Pregnancy (or willing to become pregnant) is NOT an exclusion criteria (unless specified in the respective satellite protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) diagnosed with cutaneous melanoma or non-melanoma skin cancer (including basal cell carcinoma and squamous cell carcinoma) who are treated at University Hospitals Leuven. Participants must provide voluntary written informed consent prior to any study-related procedures. Patients unable or unwilling to provide consent are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2050-01 (Estimated); Study Completion 2051-01 (Estimated)

PRIMARY OUTCOMES:
Establishment of a biobank of human body material (HBM) and clinical data | Baseline (diagnosis and informed consent) through study completion, approximately 10 years.
  Successful prospective collection and long-term storage of blood (serum, plasma, DNA), tissue samples, and associated clinical data from patients with cutaneous melanoma and non-melanoma skin cancer.

SECONDARY OUTCOMES:
Availability of biobank resources for future research | Baseline (diagnosis and informed consent) through study completion, approximately 10 years.
  Number of approved satellite protocols using biobank samples and data for translational research.

CONTACTS AND LOCATIONS:
Locations (1):
- UZLeuven, Department of Dermatology, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly. This study is an umbrella protocol for the collection and long-term storage of human body material (HBM) and associated clinical data in a biobank. Data are pseudonymized and linked to biological samples for future research projects, which require separate ethical approval. Access to IPD will only be granted under strict conditions through approved satellite protocols and in compliance with GDPR and Belgian privacy laws.